CLINICAL TRIAL: NCT07024381
Title: The Predictive Value of Heart Rate Variability for the Prognosis of Patients With Mild to Moderate Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Peng Yang (Other)
Responsible Party: Sponsor-Investigator, Peng Yang, phd., The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Other Study IDs: 2024-712
Record Dates: First submitted 2025-05-13; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: TBI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This study takes the GOS score at 6 months follow-up after patient discharge as the primary endpoint

SUMMARY:
This study adopts a retrospective design, continuously including patients with TBI treated at the Emergency Trauma Center of the First Affiliated Hospital of Suzhou University from May 2017 to September 2024. Investigators used the hospital's electronic medical record system to collect clinical data. The patients' age, gender, history of diabetes, history of hypertension, medication history, mechanism of injury, mean arterial pressure, Glasgow Coma Scale, and other information were recorded upon emergency admission. Laboratory indicators included white blood cell count, hemoglobin (HB) levels, platelet count, C-reactive protein, international normalized ratio (INR), and albumin. Myocardial injury markers included alpha-hydroxybutyrate dehydrogenase, creatine kinase, lactate dehydrogenase, aspartate aminotransferase, creatine kinase-MB (CK-MB), myoglobin, NT-pro BNP, and high-sensitivity troponin T. Additionally, continuous ECG monitoring was conducted for 24 hours after admission.

DETAILED DESCRIPTION:
This study adopts a retrospective design, continuously including patients with TBI treated at the Emergency Trauma Center of the First Affiliated Hospital of Suzhou University from May 2017 to September 2024. Investigators used the hospital's electronic medical record system to collect clinical data. The patients' age, gender, history of diabetes, history of hypertension, medication history, mechanism of injury, mean arterial pressure, Glasgow Coma Scale, and other information were recorded upon emergency admission. Laboratory indicators included white blood cell count, hemoglobin (HB) levels, platelet count, C-reactive protein, international normalized ratio (INR), and albumin. Myocardial injury markers included alpha-hydroxybutyrate dehydrogenase, creatine kinase, lactate dehydrogenase, aspartate aminotransferase, creatine kinase-MB (CK-MB), myoglobin, NT-pro BNP, and high-sensitivity troponin T. Additionally, continuous ECG monitoring was conducted for 24 hours after admission.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of traumatic brain injury
2. GCS score between 9-15;
3. Head and neck simplified injury score (AIS) ≤4;

Exclusion Criteria:

1. clinical diagnosis of tumors, active infections, or hematologic diseases;
2. those who have received treatment with beta-blockers, anticholinergic drugs, or anticoagulants within 6 months before admission;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild-to-moderate TBI patients admitted to our emergency department (May 2017- Sep 2024) were diagnosed by CT, symptoms, history, and physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Score | 6 months after discharge
  Glasgow Outcome Score
  1. Dead: As a direct result of brain trauma, or due to secondary complications, or other complications
  2. Vegetative State: Patients who remain unresponsive and speechless…. 3， Severe Disability: The patient is conscious but needs the assistance of another person for some activities of daily living every day 4， Moderate Disability: Such a patient can look after himself at home, get out and about to the shops, and travel by public transport. However, some previous activities, either at work or in social life, are now no longer possible because of either physical or mental deficit 5， Good Recovery: This indicates the capacity to resume normal occupational and social activities, although minor physical or mental deficits may exist. Social outcomes should be included in the assessment here, such as leisure activities and family relationships.
Standard deviation of all NN intervals（SDNN） | Day 1 post-TBI.
  This metric measures the standard deviation of normal beat-to-beat intervals (SDNN) present within the heart rhythm. It is a time domain measure of heart rate variability（HRV）, and it serves as a marker of overall adaptability of the nervous system.
The average of all 5-minute standard deviations of NN intervals across a 24-hour period (SDNN index) | day 1 post TBI
  The average of all 5-minute standard deviations of NN intervals across 24 hours (SDNN index). Reflects combined parasympathetic and sympathetic modulation
The root mean square of successive differences between NN intervals (RMSSD) | Day 1 post-TBI
  The Root Mean Square of Successive Differences between NN intervals (RMSSD) quantifies the variability in time intervals between consecutive normal heartbeats (NN intervals) on an electrocardiogram (ECG). Reflects parasympathetic (vagal) tone, as it captures rapid, beat-to-beat changes in heart rate mediated by the autonomic nervous system. A higher RMSSD indicates greater HRV and adaptability of the cardiovascular system, often associated with better stress resilience and recovery.
The proportion of consecutive NN intervals differing by over 50 ms, relative to the total number of NN intervals (pNN50) | day 1 post-TBI
  A higher pNN50 indicates greater parasympathetic dominance. A lower pNN50 suggests reduced vagal tone, common in stress, aging, or pathologies.
Triangle index | day 1 post TBI
  The Triangle Index is a global measure of heart rate variability derived from the geometric properties of an NN interval histogram. A higher value indicates greater overall HRV, reflecting healthy autonomic nervous system function.
HRV High Frequency Power | Day 1 post-TBI
  Baseline level of High Frequency HRV power (0.15-0.4 Hz) measured in ms2/Hz recorded on day 1 of TBI
HRV low frequency power | Day 1 post- TBI
  Low-frequency (LF) power (typically 0.04-0.15 Hz) is a spectral component of HRV reflecting mixed sympathetic and parasympathetic influences on heart rate, with potential contributions from baroreflex activity.
HRV very low frequency power | Day 1 post- TBI
  VLF (Very-Low-Frequency) power is a spectral component of heart rate variability (HRV) in the 0.0033-0.04 Hz range (or sometimes <0.05 Hz). VLF is linked to long-term autonomic and neurohormonal control.

SECONDARY OUTCOMES:
Glasgow Coma Scale | On Day 1 after TBI onset
  Its values range from 3 to 15. 13 to 15: Mild traumatic brain injury (mTBI). 9 to 12: Moderate TBI.3 to 8: Severe TBI.
Hypertension history | On Day 1 after TBI onset
Diabetes history | On Day 1 after TBI onset
Age | Baseline
White Blood Cell Count | On Day 1 after TBI onset
  White Blood Cell (WBC) count refers to the measurement of the total number of white blood cells (leukocytes) per microliter (µL) or cubic millimeter (mm³) of blood. These cells are a crucial component of the immune system, playing essential roles in defending the body against infections, foreign substances, and diseases.
Hemoglobin | On Day 1 after TBI onset
  Hemoglobin (Hb or Hgb) is an iron-containing protein found in red blood cells (RBCs) that binds oxygen in the lungs and delivers it to tissues throughout the body while also transporting carbon dioxide back to the lungs for exhalation.
Platelets (thrombocytes) | On Day 1 after TBI onset
  Platelets (thrombocytes) are small, colorless cell fragments in the blood that play a crucial role in clotting and stopping bleeding. The platelet count (PLT) measures the number of platelets per microliter (μL) of blood.
C-Reactive Protein (CRP) | On Day 1 after TBI onset
  C-reactive protein (CRP) is a liver-produced protein that increases rapidly in response to inflammation, infection, or tissue damage. It is a key acute-phase reactant used to detect and monitor inflammatory conditions.
International Normalized Ratio | On Day 1 after TBI onset
Albumin | On Day 1 after TBI onset
Alpha-Hydroxybutyrate Dehydrogenase | On Day 1 after TBI onset
Creatine Kinase | On Day 1 after TBI onset
Lactate Dehydrogenase | On Day 1 after TBI onset
Aspartate Aminotransferase | On Day 1 after TBI onset
Creatine Kinase-MB | On Day 1 after TBI onset
Myoglobin | On Day 1 after TBI onset
N-Terminal pro-BNP | On Day 1 after TBI onset
High-Sensitivity Troponin T | On Day 1 after TBI onset

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine，the First Affiliated Hospital of Soochow University., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Publish in the form of an academic paper

REFERENCES:
- [Derived] Wu C, Liu L, Chen D, Zhu W, Xu F, Yang P. The Predictive Value of Heart Rate Variability for the Prognosis of Patients with Mild to Moderate Traumatic Brain Injury. Neurol Ther. 2025 Oct;14(5):1889-1901. doi: 10.1007/s40120-025-00792-0. Epub 2025 Jul 4. PMID 40614040